CLINICAL TRIAL: NCT04568395
Title: Acute Impact of Switching From Tobacco Cigarettes to E-Cigarettes in People Living With HIV
Brief Title: Acute Effects of TCIG vs ECIG in PLWH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-001179
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: E Cigarette Use; Vaping; Smoking; Tobacco Smoking; Nicotine Use Disorder; Qt Interval, Variation in; HIV I Infection; Oxidative Stress; Inflammation
MeSH Terms: conditions — Vaping; Smoking; Tobacco Smoking; Tobacco Use Disorder; Inflammation

STUDY DESIGN:
Intervention Model Description: Crossover with 1 week washout
Masking Description: single (outcomes assessor) code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLWH smoker (Experimental): PLWH who smoke will undergo 3 interventions : acute TCIG use, acute ECIG use and acute sham control
  Interventions: Other: TCIG; Other: ECIG; Other: sham control

INTERVENTIONS:
Other: TCIG — Use a TCIG
Other: ECIG — Use an ECIG
Other: sham control — Use a sham control (empty ECIG)

SUMMARY:
Randomized controlled trial of acute use of electronic cigarette or tobacco cigarette on parameters of ventricular repolarization and inflammation/oxidative stress.

DETAILED DESCRIPTION:
On separate days, participants will undergo 3 different exposures: an acute e-cigarette exposure, an acute tobacco cigarette exposure, and a sham (empty e-cigarette) control . Before and after the acute exposure, participants will have blood drawn for inflammation/oxidative stress markers and undergo a 5-minute ECG recording.

ELIGIBILITY:
Inclusion Criteria:

Chronic (> 1year) TCIG smoker HIV positive Stable ART Viral count non-detectable CD4 >500

Exclusion Criteria:

Known major illness (heart disease, diabetes, lung or liver disease) Daily recreational drug use, including cannabis >2 alcoholic drinks per day Obesity (>30 kg/m2) Recent (<3 months) infection

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Tpe | Change in Tpe 5 minutes after cigarette use
  interval indicative of ventricular repolarization measured on ECG
Tpe/QT | Change in Tpe/QT after cigarette use
  interval indicative of ventricular repolarization measured on ECG
Tpe/QTc | Change in Tpe/QTc after cigarette use
  interval indicative of ventricular repolarization measured on ECG
Total Cellular Reactive Oxygen Stress | within 4 hours of cigarette use
  total cellular oxidative stress measured by flow cytometry

SECONDARY OUTCOMES:
QT | Change in QT after cigarette use
  interval indicative of ventricular repolarization measured on ECG
QTc | Change in QTc after cigarette use
  interval indicative of ventricular repolarization measured on ECG

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - UCaliforniaLA, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No